CLINICAL TRIAL: NCT00001195
Title: Endocrine Studies of Healthy Children
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 840169; 84-CH-0169
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2014-10-20

CONDITIONS: Healthy
Keywords: Development; Hormones; Growth; Metabolism; Eating Behavior; Body Composition; Normal Volunteer
MeSH Terms: conditions — Feeding Behavior

SUMMARY:
Researchers would like to determine normal ranges for hormone levels and to learn more about the genetics involved in hormone production and action. Researchers will take samples of blood, urine, saliva, and stool from healthy children ages 5-17 in order to study different aspects of hormones.

Establishing a range of normal hormone levels in children will make diagnosing illnesses with abnormal levels of hormones much easier. Hormone levels in the body can change throughout the day. By collecting samples at different times researchers hope to learn more about the normal daytime and nighttime patterns of hormone secretion. Because some hormone levels change with body size, researchers will also take measurements of patient's body composition.

This study will involve children and observe them as inpatients or as outpatients. <TAB>

DETAILED DESCRIPTION:
We wish to obtain blood, urine, saliva, and stool specimens from healthy children ages 2-18 years for use in establishing the normal ranges of levels of hormones and the variations in genes that are important for hormones to act. Such hormone values are extremely important to allow endocrinologists to determine when hormone levels are truly abnormal in children suspected of an illness. Because the values of some hormones change with body size, we will obtain measurements of body composition when studying such hormones. Children participating in this study may be studied in the outpatient clinic (at most 2 blood draws) or as inpatients on the pediatric ward (for frequent blood sampling using an intravenous line over a 24-hour period). Other studies that may be performed as part of this study include ultrasound examinations of the thyroid, adrenal, ovaries or testes, and x-ray of the hand and wrist for bone age determination.

ELIGIBILITY:
* INCLUSION CRITERIA:

Good general health.

Age 2 to 18 years.

EXCLUSION CRITERIA:

Volunteers will be excluded for the following reasons:

Presence of renal, hepatic, gastrointestinal, most endocrinologic (e.g., Cushing's syndrome) or pulmonary disorders (other than asthma not requiring continuous medication);

Individuals who have, or whose parent or guardians have, current substance abuse or a psychiatric disorder or other condition which, in the opinion of the investigators, would impede the ability to give informed consent or possibly hinder completion of the study;

Subjects who regularly use prescription medications are not eligible. The use of over-the-counter medications will be reviewed on a case-by-case basis;

For those sub-studies involving MRI, inability to undergo MRI (e.g., volunteers with metal within their bodies including cardiac pacemakers, neural pacemakers, aneurysmal clips, shrapnel, ocular foreign bodies, cochlear implants, non-detachable electronic or electromechanical devices such as infusion pumps, nerve stimulators, bone growth stimulators, etc. that are contraindications).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1247 (Actual)
Dates: Start 1984-08-28; Study Completion 2014-10-20

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nisula BC, Loriaux DL, Wilson YA. Solid phase method for measurement of the binding capacity of testosterone-estradiol binding globulin in human serum. Steroids. 1978 May;31(5):681-90. doi: 10.1016/s0039-128x(78)80008-7. No abstract available. PMID 566971
- [Background] Nisula BC, Dunn JF. Measurement of the testosterone binding parameters for both testosterone-estradiol binding globulin and albumin in individual serum samples. Steroids. 1979 Dec;34(7):771-91. doi: 10.1016/0039-128x(79)90090-4. PMID 575443
- [Background] Wehmann RE, Rubenstein HA, Nisula BC. A sensitive, convenient radioimmunoassay procedure which demonstrates that serum hTSH is suppressed below the normal range in thyrotoxic patients. Endocr Res Commun. 1979;6(3):249-55. doi: 10.3109/07435807909061799. PMID 520279
- [Derived] Han JC, Reyes-Capo DP, Liu CY, Reynolds JC, Turkbey E, Turkbey IB, Bryant J, Marshall JD, Naggert JK, Gahl WA, Yanovski JA, Gunay-Aygun M. Comprehensive Endocrine-Metabolic Evaluation of Patients With Alstrom Syndrome Compared With BMI-Matched Controls. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2707-2719. doi: 10.1210/jc.2018-00496. PMID 29718281
- [Derived] Radin RM, Tanofsky-Kraff M, Shomaker LB, Kelly NR, Pickworth CK, Shank LM, Altschul AM, Brady SM, Demidowich AP, Yanovski SZ, Hubbard VS, Yanovski JA. Metabolic characteristics of youth with loss of control eating. Eat Behav. 2015 Dec;19:86-9. doi: 10.1016/j.eatbeh.2015.07.002. Epub 2015 Jul 18. PMID 26210388
- [Derived] Tanofsky-Kraff M, Shomaker LB, Stern EA, Miller R, Sebring N, Dellavalle D, Yanovski SZ, Hubbard VS, Yanovski JA. Children's binge eating and development of metabolic syndrome. Int J Obes (Lond). 2012 Jul;36(7):956-62. doi: 10.1038/ijo.2011.259. Epub 2012 Jan 10. PMID 22234282